CLINICAL TRIAL: NCT06133036
Title: Fecal Continence Outcomes and Quality of Life After Excision of Sacrococcygeal Teratma (Retrospective Study)
Brief Title: Fecal Continence Outcomes and Quality of Life After Excision of Sacrococcygeal Teratoma (Retrospective Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Kamal Mohamed Sayed Khalil, resident-pediatric surgery department, Sohag University
Other Study IDs: Soh-Med-23-10-10MS
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Sacrococcygeal Teratoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sacrococcygeal teratoma is one of the most common tumors that occur in the neonatal period. It presents either as a mass protruding from the sacrococcygeal region or as a pelviabdominal mass according to the type. Surgical excision is the main treatment, most masses are benign, however some are malignant and require radiotherapy or chemotherapy. Complications may occur due to pressure resulting from the tumor growth in the fetal period, or due to damage to important near tissues during surgical excision. Postoperative complications may be urinary as neurogenic bladder, Lower gastrointestinal as constipation, soiling or incontinence. In this work we study the outcomes of fecal continence through a questionnaire and its effect on the quality of life of the affected children.

ELIGIBILITY:
Inclusion Criteria:

* all patients with sacrococcygeal teratoma operated after july 2010 and older than 3 years old.

Exclusion Criteria:

* Patients lost to follow up before 6 months after surgery.
* Patients with Currarino triad.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients operated in Sohag university hospital after july 2010 for sacrococcygeal teratoma.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Fecal continence | 6 months
  Measured by Rintala continence score

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided